





## **Informed Consent Form (ICF)**

## **Lung Immune Challenge Study:**

Controlled Exposure to Inhaled Resiquimod (R848) to Study Mechanisms of Inflammation

| Participant name | | | |
|---|---|---|---|
| Study ID | | | |
| <u>'</u> | | | Please<br>initial |
| I confirm that I have read the Participant Information Sheet (version 1.0 dated 19.04.24). I have had the opportunity to consider the information, ask questions and had these answered satisfactorily. | | | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| I understand that tissue and any cells derived from my samples will be analysed including for genes and gene activity and may be cultured and stored in the long term. I agree that stored cells and tissue may be shared with third party academic or industrial partners in the United Kingdom or abroad for medical research purposes only. | | | |
| I give permission for relevant sections of my medical notes and information collected during the study to be looked at may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. | | | |
| I agree that my personal and clinical data can be shared with third party colleagues for scientific related research purposes. I understand this information will <u>not</u> include any personal identifying details that would allow me to be identified by a third party. | | | |
| I agree that if required my general practitioner (GP) may be informed of my participation in the study, including any necessary exchange of information about me between my GP and the research team. | | | |
| I agree to take part in the current study | | | |
| Optional: I agree to be contacted about future research studies although I am not obliged to take part. | | | |
| Name of Participant | Date | Signature | |
| Name of Person taking<br>Consent | g Date | Signature | |

Lung Immune Challenge Study ICF, 19.04.24, Version 1.0, IRAS project ID: 340091